CLINICAL TRIAL: NCT06415435
Title: A Multi-Center, Open-Label, Prospective Study of the Sylfirm X Device for the Treatment of Melasma
Brief Title: Sylfirm X Radiofrequency Microneedling for the Treatment of Melasma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benev Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIOL-MEL-2022
Record Dates: First submitted 2024-04-30; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sylfirm X Treatment with Sunscreen (Experimental)
  Interventions: Device: Radiofrequency Microneedling
- No Treatment, Sunscreen Only (No Intervention)

INTERVENTIONS:
Device: Radiofrequency Microneedling — Sylfirm X radiofrequency microneedling device
  Arms: Sylfirm X Treatment with Sunscreen

SUMMARY:
Microneedling radiofrequency technology has been shown in clinical studies to improve skin quality, tone, pigment, and to treat various skin conditions related to aging.

The purpose of this study is to evaluate efficacy and safety of Sylfrim X device for the treatment of melasma.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to read, understand and sign informed consent form.
2. Healthy females, 19 and older
3. Fitzpatrick I-VI
4. Has melasma
5. Willing to have RF microneedling treatment and able to adhere to treatments, follow up schedule, and post-treatment instructions
6. Willing to have limited sun exposure and use sunscreen on treatment area everyday for duration of study
7. Willing to have photographs taken of treatment area and agree to use of photographs
8. Willing to refrain from using topical corticosteroids, or retinoids
9. Agree to undergo procedure in treatment area during study
10. Females: not pregnant, or lactating and is either post-menopausal, surgically sterilized, or using birth control at least 1 month prior to enrollment
11. Willing to wear sunscreen and apply once daily in morning and every 2 hours

Exclusion Criteria:

1. Participation in a clinical trial of another drug, or device administered to the treatment area, within 3 months prior to enrollment or during the study.
2. Any type of prior cosmetic treatment to the target area within 3 months of study participation, such as laser/light procedures, and those used for general aesthetic correction, neuromodulators, facial peel, lightening creams, or facial surgery.
3. Any fillers within 3 months prior to enrollment or during the study.
4. Use of prescription topicals in the treatment area within one month prior to treatment or use of topical agents one week prior to treatment that may cause facial sensitivity.
5. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including but not limited to, open lacerations or abrasions, hidradenitis, rash, infection, or dermatitis of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion).
6. . Pregnant and/or breastfeeding or planning to become pregnant.
7. Significant concurrent illness, such as diabetes mellitus, immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or using immunosuppressive medication.
8. Any use of any medication that is known to increase sensitivity to light or hypersensitivity to light exposure according to the Investigator's discretion.
9. History of keloid scarring, hypertrophic scarring or abnormal wound healing or prone to bruising.
10. If you have a history of squamous cell carcinoma or melanoma in the treatment area, this includes basal cell carcinoma unless: basal cell carcinoma was treated or excised with no evidence of reoccurrence within the past 6 months prior to screening. Squamous cell carcinoma in situ, which has been treated or excised without evidence or reoccurrence within the past 6 months prior to screening.
11. . History of epidermal or dermal disorders (particularly if involving collagen or micro vascularity), including collagen vascular disease or vasculitis disorders.
12. A history or active skin condition that in the opinion of the Investigator may interfere/confound with the treatment.
13. History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.

    Sponsor: VIOL Version 1, 25APR2022 Protocol: VIOL-MEL-2022 Page 18 of 47
14. History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
15. Excessively tanned or active sun tan in facial area to be treated, or unable/unlikely to refrain from tanning during the study.
16. Excessive facial hair in the area to be treated (beards, sideburns, and/or mustache,) that would interfere with diagnosis, assessment, and treatment.
17. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study, including excessive alcohol or drug abuses, or a condition that would compromise the subject's ability to comply with the study requirements.
18. To reduce potential effects of hormonal changes in melasma, a 6-month washout period is required for female subjects who have recently stopped or started contraceptive use, have recently delivered an infant, or have stopped breastfeeding.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of photos accurately identified as post-treatment photo vs. baseline by a blind investigator from 0-100% | 28 days
  Success criteria: 80% accuracy in identifying the baseline photo from post-treatment photos.

SECONDARY OUTCOMES:
Change in Modified Melasma Area and Severity Index (mMASI) scale measured by investigator (range 0-24), a lower score indicating clearer skin. | 28 days
  The Modified Melasma Area and Severity Index scale will be utilized to grade melasma severity. Success criteria: improvement by 1 point, ie. at least 1 point lower than baseline.
Percentage of subjects with an increase in satisfaction level assessed from Melasma Quality of Life questionnaire (MELQoL) after treatment compared to baseline | 28 days
  MELQoL is a questionnaire on a scale of 0 to 7 on how the patients feel about skin appearance, skin condition, embarrassment about skin condition, etc.
Statistical improvement of investigator Global Aesthetic Improvement Scale (GAIS) | 28 days
  Success criteria: On a scale of -1 (skin got worse) to 3 (skin very much improved), incidence of subject improvement was statistically significant.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Scripps Health, La Jolla, California
  - Dermatology, Laser & Vein Specialists of the Carolinas, PLLC, Charlotte, North Carolina
  - Refresh Dermatology, Houston, Texas